CLINICAL TRIAL: NCT07311382
Title: Effect of Administering an Oil Prepared at CIAL as a Means to Supply Long-chain Fatty Acids to Very Preterm Newborns
Brief Title: Effect Partial Digested Triglycerides on Supply Long-chain Fatty Acids to Very Preterm Newborns
Acronym: DHA-CIAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Miguel Saenz de Pipaon, MD, Hospital Universitario La Paz
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: HULP-6548
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Plasma Concentration
Keywords: carbon isotopes; Fatty Acids; Phospholipids; Long growth

STUDY DESIGN:
Intervention Model Description: One arm adminitration of ARA and DHA 160 / 80 mg/kg/day vs standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARA: DHA supplementation (Experimental): Experimental group will receive supplementation with fatty acids, ARA and DHA 160 and 80 mg/kg/day respectively. It will begin once consent is obtained and will continue until discharge or 36 weeks, whichever comes first.
  Interventions: Dietary Supplement: Measure long-chain fatty acids in plasma after administration of a supplement from the first days of life until 36 weeks postmenstrual age
- Control (No Intervention): Usual care

INTERVENTIONS:
Dietary Supplement: Measure long-chain fatty acids in plasma after administration of a supplement from the first days of life until 36 weeks postmenstrual age — Long-chain fatty acids in plasma after administration of a supplement from the first days of life until 36 weeks postmenstrual age
  Arms: ARA: DHA supplementation

SUMMARY:
Main objective: To determine the bioavailability of long-chain fatty acids in very preterm newborns after administering a supplement from the first days of life until 36 weeks postmenstrual age compared to children who did not receive the supplement.

The primary variable will be assessed by measuring the increase in the proportion of docosahexaenoic acid and arachidonic acid in plasma phospholipids. 1 ml of the milk received by the child will be collected to evaluate fatty acid intake naturally at 10, 21 days, and 36 weeks postmenstrual age. Stool samples from the child will also be collected at all time points to evaluate the elimination of the supplement.

Secondary objectives: 1. Determine the influence of different polymorphisms (SNPs) on the proportion of fatty acids in plasma phospholipids at birth and after the intervention. This will be evaluated through the analysis of genes related to fatty acid metabolism in buccal mucosa cells. 2. Determine the effect of supplementation on: • Changes in the microbiota from birth to the end of the intervention. • Maturation of brain function. • Brain size. • Lung development. • Growth. Evaluated through: • Metataxonomics • Amplitude-integrated electroencephalography (aEEG) at 34 weeks postmenstrual age (PMA). One channel (P3-P4). aEEG traces were recorded for at least 4 hours using the NicoletOne® EEG system monitor (Natus Medical Inc., CA, United States). The tracings will be evaluated following the maturation scoring system developed by Burdjalov et al.

* Cranial ultrasounds (cUS) will be performed at 36 weeks PMA (Canon R, Aplio 500; transducer set at 8-10 MHz). All linear measurements on cUS will be blinded. cUS measurements will be obtained in the following planes:

  * mid-coronal plane at the level of the foramina of Monro (anterior horn width, ventricular index, ventricle-to-brain ratio, frontal white matter height, interhemispheric fissure and subarachnoid space, coronal atrial plane [ventricular width at midbody]),
  * mid-sagittal plane (corpus callosum width and length, corpus callosum-fastigium length, vermis height and A-P width),
  * parasagittal plane through the lateral ventricles (thalamo-occipital distance of the lateral ventricles), and
  * mastoid view (coronal transverse cerebellar diameter). The following cUS variables will be collected: intraventricular hemorrhage, post-hemorrhagic ventriculomegaly, cerebellar hemorrhage, and white matter injury.
* Respiratory severity was also assessed using the SatO2/FiO2 ratio, the non-invasive pulse oximetry ratio SatO2/FiO2 which estimates the PaO2/FiO2 ratio, or between peripheral oxygen saturation by pulse oximetry (Nellcor™ SpO₂ bedside monitoring system, PM100N, (Covidien, Boulder, Colorado, USA)) and the fraction of inspired oxygen (FiO2, via ventilator, CPAP devices, or oximeters).

  * Birth weight (g), length (cm), and head circumference (HC, cm) will be recorded at birth, 21 days, and 36 PMA at discharge.
  * Z-scores will be calculated using the revised Fenton growth charts.
  * The Z-score difference between 36 weeks and birth will be calculated for weight, length, and HC.
  * Additionally, growth velocity will be calculated using the following equation:

Weight velocity is reported as g/kg/day and length and HC as cm/day Weight velocity = (1000 * Ln (Weight at 36 PMA / birth weight)) / Number of days Length and HC velocity = (Length or HC at 36 PMA / Length or HC at birth) / Number of days

Safety: To monitor patients' well-being in this study, the following will be performed:

* Risk of adverse events and serious adverse events.
* Medication use
* Complete blood count Design: One arm, comparison with controls recruited in the recently completed Mead Johnson study. Enrolled children will receive supplementation with fatty acids, ARA and DHA at 160 and 80 mg/kg/day, respectively. It will start once consent is obtained and continue until discharge or 36 weeks, whichever comes first.

Study product: Product of enzymatic glycerolysis of arachidonic acid oil and microalgae oil. Product fatty acid profile in %: Arachidonic 20:4 35.94; DHA C22:6 18.17.

Study population: Preterm newborns under 32 weeks of gestational age at birth. Inclusion criteria:- Informed consent, < 32 weeks of gestational age Duration of intervention: Until discharge or 36 weeks, whichever occurs first. Sample size: n = 15 has been established according to previous results from a study with similar characteristics and with the studies conducted in the two projects funding this study.

Analysis: The increase in the percentage of polyunsaturated fatty acids in plasma phospholipids from birth to week 36 will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborns less than 32 weeks of gestational age at birth.
* Informed consent accepted

Exclusion Criteria:

* Not cord blood available

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
DHA and AA in plasma | From birth to 36 weeks PMA
  The increase in the proportion of docosahexaenoic acid and arachidonic acid in plasma phospholipids.

CONTACTS AND LOCATIONS:
Locations (1):
- La Paz Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No